CLINICAL TRIAL: NCT00302991
Title: Quality of Life and Adverse Effects in Epilepsy Patients According to Treatment Group (EPIKA)
Brief Title: Quality of Life and Adverse Effects in Epilepsy Patients (EPIKA)
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Other Study IDs: N01247; EPIKA
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Epilepsy
Keywords: Observational; cross-sectional; health-related quality of life; adverse effects; Baker´s AEP scale validation; epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational, multicentre, epidemiological study to determine the HRQOL of patients with epilepsy according to treatment sub-group and to validate the Spanish version of the Adverse Events Profile, produced by G. Baker et al. Three treatment groups will be examined: patients receiving only a new anti-epilepsy drug (AED), patients receiving a "classic" AED; patients receiving combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Epileptic adult patients treated at a stable dose with one or more AEDs for ≥ 3 months

Exclusion Criteria:

* Symptomatic epilepsy due to malignant brain tumour or progressive brain disease.
* Confirmed diagnosis of a concomitant chronic disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial M. Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Barcelona, Spain